CLINICAL TRIAL: NCT03445715
Title: A Single Dose Clinical Trial to Study the Safety of ART-I02 in Patients With Rheumatoid Arthritis
Brief Title: ART-I02 in Patients With Rheumatoid Arthritis With Inflamed Wrists
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arthrogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART-I02-001
Record Dates: First submitted 2018-02-01; First posted 2018-02-26 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort I (Experimental): Single intra-articular injection ART-I02: 2.4x10E12 vg / wrist joint
  Interventions: Genetic: ART-I02
- Cohort II (Experimental): Single intra-articular injection of ART-I02: 2.4x10E13 vg / wrist joint
  Interventions: Genetic: ART-I02
- Cohort III (Experimental): Single intra-articular injection in the wrist joint of ART-I02 Maximum Tolerated Dose (MTD) as assessed in cohorts I and II:
  Interventions: Genetic: ART-I02

INTERVENTIONS:
Genetic: ART-I02 — Single Intra-articular injection in the wrist joint
  Other Names: Recombinant AAV type2/5 containing a hIFN-b gene

SUMMARY:
This study will evaluate the safety and tolerability of a single intra-articular administration of ART-I02 (AAV5.NF-kB.IFN-β), a recombinant adeno-associated virus (AAV) type 5 vector in subjects with RA and active arthritis of a wrist.

DETAILED DESCRIPTION:
DMARDs such as methotrexate, sulfasalazine and leflunomide used alone or in combination, are considered to be standard treatment for RA and may be combined with other conventional DMARDs and/or corticosteroids and/or anti-inflammatory or centrally working analgetics (NSAIDS). During the last decade, treatment with biological (e.g. TNF-inhibitors), together with improved timing and dosing of conventional therapy, has significantly improved the outcome in a significant proportion of RA patients. The advent of biologicals and implementation of more intensive treatment protocols has significantly improved the outcome in a significant proportion of RA patients and prevented disabilities. However, drug-free remissions are still rare and hence most RA patients require continued immunosuppressive treatment which predisposes them to potentially serious infections. Also up to 50% of RA patients continue to suffer from symptomatic disease. Intra-articular glucocorticoids are often used in these patients, e.g. when single joints are inflamed. The duration of their effect is however variable. It regularly occurs in clinical practice that reasonable clinical remission in rheumatoid arthritis patients is achieved with current treatment options, but that one or more joints still display persistent signs of inflammation while the inflammation of other joints has been greatly reduced. This means that for the joint(s) still affected by active inflammation other therapies are required.

There is a need for additional RA therapies with good tolerability and efficacy profiles that can be used in patients who suffer from a few inflamed joints despite previous treatment. Intra-articular gene therapy could provide a solution by providing local treatment for arthritis, with prolonged expression of a therapeutic protein at the site of inflammation after a single injection.

ART-I02 is an investigational new drug, expressing human IFN-β from a recombinant (r) adeno-associated virus type 5 (rAAV5) β under the influence of a promoter, which is induced by an inflammatory stimulus. Due to the relapsing nature of RA, therapeutic expression should be maximal during flare-ups of the disease. This is achieved by employing the NF-kB responsive promotor to regulate expression of IFN-β. Under inflammatory conditions, the NF-kB responsive promoter will be activated in the synovium and will upregulate the expression of hIFN-β and turned down during remission. In this way, transgene expression can be controlled, following the intermittent course of disease. The selection of IFN-Beta as the therapeutic protein is based on the notion that IFN-β has anti-inflammatory, and bone and cartilage protective effects, which have been extensively demonstrated in non-clinical studies.

This is a phase I open label, dose escalating study to investigate the safety of a single intra-articular ART-I02 injection in patients with RA and active arthritis of a wrist.

In a two-phase staggered dose escalation design, dosing will start with a low dose (2.4x1012 vg/ wrist) and progress to the highest dose of 2.4x1013 vg/wrist. Three patients will be enrolled at each of the two dose levels. The interval between dosing of patients within dose escalation cohorts I and II is at least two weeks to allow for safety evaluation by the investigator. Following dosing of the last patient in cohort I and II, a dosing pause of two weeks is included to allow an assessment of the safety data by the Data Review Committee (DRC). Enrollment in the subsequent cohort will continue only after a thorough assessment of safety and tolerability data (medical history, vital signs, physical examination, laboratory parameters and adverse events) through day 14 post dose; for the first treated patient in each cohort safety data up to a minimum of six weeks, for the second patient up to a minimum of four weeks and for the third patient up to a minimum of two weeks are available at the time of the assessment of the safety data by the DRC. In cohort III nine patients will be administered the highest safety dose of ARTI02 as determined in the previous dose escalating cohorts (cohorts I and II) and following a thorough assessment of all available safety data including a minimum of 2 weeks data post ART-I02 administration from the 3rd patient of cohort II. The interval between dosing of patients within cohort III is at least one week. Cohort III is added to the study to substantiate the safety profile of the highest tolerated dose of ART-I02. The consideration to treat one joint in this clinical study is that it provides the opportunity to examine the administration of a single dose at the site where the promoter is activated and where the therapeutic protein IFN-β is required.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with RA aged ≥18 years.
2. Patient has been diagnosed with RA according to the 2010 American College of Rheumatology/ European league against rheumatism (ACR/EULAR) criteria for the classification of RA, outlined in appendix A.
3. Inflammation of the target wrist due to active RA as confirmed by MRI, and the (symptoms of) inflammation is (are) not satisfactorily controlled by current best-standard therapy, and/or that the patient could benefit from better therapeutic efficacy, according to judgment of the investigator.
4. Written informed consent, able and willing to comply with the requirements of the study protocol.
5. Judged to be in general good health with, in the opinion of the investigator, no other clinically significant and relevant abnormalities of medical history, and no abnormalities at the physical examination, vital signs, electrocardiography (ECG) and laboratory safety tests, performed at the screening visit and/or prior to administration of ART-I02.
6. Females are not pregnant nor lactating.
7. All male patients use effective contraception in combination with barrier contraception until three consecutive semen samples are negative for ART-I02 genomic DNA. All female patients of childbearing potential use effective contraception in combination with barrier contraception for the first three months after administration.

Exclusion Criteria:

1. Arthrodesis or joint replacement of the target wrist prior to inclusion.
2. Known hypersensitivity to natural or recombinant hIFN-β, or to any excipients.
3. Contra-indication for intra-articular treatment.
4. Presence of neutralizing antibody (Nab) titers against adeno-associated virus type 5 (AAV5) and/or hIFN-β.
5. Active infectious disease of any nature, including clinical active viral infections.
6. Previous treatment with an AAV 5 vector.
7. Poor functional status, defined as being bed-bound or wheelchair-bound.
8. Intra-articular corticosteroid treatment within one month prior to administration of the study medication.
9. Participation in an investigational drug or device study within 90 days prior to screening or more than 4 times per year.
10. Positive for human immunodeficiency virus (HIV) infection, hepatitis C antibodies or hepatitis B surface antigen.
11. Positive for anti-double-stranded DNA antibodies (dsDNA).
12. History of liver function abnormality requiring treatment, drug induced liver injury, chronic liver disease, excessive alcohol consumption or chronic alcohol induced disease.
13. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 x upper limit of normal (ULN), or bilirubin > 2 x ULN. If a patient has AST or ALT > 2 x ULN but < 2.5 x ULN, re-assessment is allowed at the investigator's discretion.
14. Severely impaired renal function (estimated glomerular filtration rate ≤ 30 mL/min according to the Cockcroft-Gault formula).
15. Patient had a major surgery, donated or lost approximately 500 mL blood within 4 months prior to the screening visit
16. Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude.
17. Serious medical disease, such as severe liver or kidney disease, uncompensated congestive heart failure, myocardial infarction within six months, unstable angina, uncontrolled hypertension, severe pulmonary disease or active asthma, demyelinating neurological disease, depression or a history of depression, history of seizures or epilepsy, uncontrolled epilepsy, or history of cancer (other than cutaneous basal and squamous cell carcinoma or cervical intraepithelial neoplasia) with less than five years documentation of a disease-free state, recurrent opportunistic infections or other concurrent medical condition that, in the opinion of the investigator, would make the patient unsuitable for the study.
18. Investigator has concerns regarding the safe participation of the patient in the trial or for any other reasons: the investigator considers the patient inappropriate for participation in the trial.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent (serious) adverse events | 5 years
  The number of and the number of patients with treatment emergent AEs will be reported by 1.treatment, MedDRA SOC and PT; 2. treatment, MedDRA SOC, PT and severity; 3.treatment, MedDRA SOC, PT and drug relatedness

SECONDARY OUTCOMES:
Change from baseline for clinical signs and symptoms of the target joint evaluated by the Composite Change Index (CCI) | Baseline, week 1, week 2 , week 4, week 8, week 12, week 16, week 20 and week 24 post administration of ART-I02
  Change from baseline of clinical signs and symptoms as measured by the aggregate score of the individual components of the CCI. Calculation of the CCI is based on changes of its components from baseline. The total CCI ranges from 0 (no effect or deterioration) to 10 (maximal effect). Successful treatment is defined as CCI ≥5.
Change from baseline after single dose of ART-I02 on overall disease activity measured by DAS28, over 24 weeks. | Baseline, week 24 post administration of ART-I02
  Change from baseline on overall disease activity measured by the DAS, a composition index measuring disease activity in RA, taking into account tenderness and swelling score of 28 joints, CRP), and general health VAS. Range of 0 to 9.4, below 3.2 low disease activity, level ≥ 3.2 active disease
Change from baseline after single dose of ART-I02 on hand function measured by Grip strength measurement in the target and contralateral joint. | Baseline, week 1, week 2 , week 4, week 8, week 12, week 16, week 20 and week 24 post administration of ART-I02
  Grip strength of the injected hand as well as the contra lateral hand is measured with the JAMAR Hydraulic Hand Dynamometer
Change from baseline after single dose of ART-I02 on hand function measured by VAS pain in the target and contralateral joint. | Baseline, week 1, week 2 , week 4, week 8, week 12, week 16, week 20 and week 24 post administration of ART-I02
  Pain in the target and contralateral joint will be assessed by a Visual Analogue Scale requiring the patient to respond by placing a vertical line on a 100-mm scale anchored at the ends by polar descriptions "no pain" and "unbearable pain".
Change from baseline after single dose of ART-I02 on hand function measured by VAS function in the target and contralateral joint. | Baseline, week 1, week 2 , week 4, week 8, week 12, week 16, week 20 and week 24 post administration of ART-I02
  Function of the target and contralateral joint will be assessed by a Visual Analogue Scale requiring the patient and physician to respond by placing a vertical lineon two separate 100-mm scales anchored at the ends by polar descriptions "no impairment" and "severe impairment
Change from baseline after single dose of ART-I02 on synovitis, bone erosion and oedema in the injected joint evaluated by MRI 12 and 24 weeks after administration of ART-I02 using the OMERACT RA MRI scoring sys | Baseline, week 12, week 24 post administration of ART-I02
  Change from baseline on synovitis and osteitis assessed by evaluating the aggregate scores of the components of the RAMRIS scoring system. Scale: 0-3 in increments of 33 % of the synovial compartment. Bone erosions will be assessed in each bone (wrists - carpal bones, distal radius, distal ulna, metacarpal bases; MCP joints - metacarpal heads, phalangeal heads) is scored separately . Scale: 0-10 in increments of 10 % of articular bone loss. Osteitis will be assessed by scoring each bone separately. Scale: 0-3 in increments of 33 % of bone oedema
Vector DNA in whole peripheral blood | Up to 24 weeks but maximally until such time that three consecutive samples have been tested negative
  Detection of vector DNA in whole peripheral blood using quantitative-PCR (Q-PCR).
Vector DNA in urine | Up to 24 weeks but maximally until such time that three consecutive samples have been tested negative
  Detection of vector DNA in urine using quantitative-PCR (Q-PCR).
Vector DNA in feces | Up to 24 weeks but maximally until such time that three consecutive samples have been tested negative
  Detection of vector DNA in feces using quantitative-PCR (Q-PCR).
Vector DNA in saliva | Up to 24 weeks but maximally until such time that three consecutive samples have been tested negative
  Detection of vector DNA in saliva using quantitative-PCR (Q-PCR).
Induction of humoral immune responses against AAV by measuring antibodies against AAV | Baseline, week 4 and week 24 post administration
  To assess immune responses against adeno-associated virus serotype 5 (AAV5) after a single intra-articular dose of ART-I02
Induction of humoral immune responses against AAV by measuring neutralizing antibodies against AAV | Baseline, week 4 and week 24 post administration
  To assess immune responses against adeno-associated virus serotype 5 (AAV5) after a single intra-articular dose of ART-I02
Induction of humoral immune responses against hIFN-β by measuring antibodies against IFN-β | Baseline, week 4 and week 24 post administration
  To assess immune responses against human interferon beta (hIFN-β) after a single intra-articular dose of ART-I02.
Induction of humoral immune responses against hIFN-β by measuring neutralizing antibodies against hIFN-β | Baseline, week 4 and week 24 post administration
  To assess immune responses against human interferon beta (hIFN-β) after a single intra-articular dose of ART-I02.
Induction of cellular immune responses against AAV5 by measuring T cell responses against AAV5 | Baseline, week 4, 8, 12, 16 and week 24 post administration
  To assess T-cell response against AAV5
Induction of cellular immune responses against hIFN-β by measuring T cell responses against hIFN-β | Baseline, week 4, 8, 12, 16 and week 24 post administration
  To assess T-cell response against hIFN-β
Effect of a single intra-articular dose of ART-I02 on inflammation markers in synovium biopsies. | Week 24
  Synovial fluid is analyzed for presence of IFN-β protein, ART-I02 vector DNA and inflammatory markers. The synovial tissue is analyzed for expression of IFN-β protein, inflammatory cytokines, proteins involved in cartilage metabolism, and histopathology and including immunohistochemical staining for cellular markers. The presence of ART-I02 vector DNA is measured.
Vector DNA in semen | Up to 24 weeks but maximally until such time that three consecutive samples have been tested negative
  Detection of vector DNA in semen using quantitative-PCR (Q-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: William O Martin, PhD, Principal Investigator — University Of Calagary
Locations (1):
- University of Calgary, Division of Rheumatology, Cumming School of Medicine, Calgary, Canada

IPD SHARING:
Plan to Share IPD: No